CLINICAL TRIAL: NCT02525016
Title: Safety Profile of IntRAvenous Lidocaine Use in Coelioscopic Bariatric Surgery
Acronym: SPIRAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL15_0057
Record Dates: First submitted 2015-08-12; First posted 2015-08-17 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Bariatric Surgery
Keywords: Bariatric surgery, lidocaine, plasmatic concentration, MonoEthylGlycineXylidide (MEGx), safety
MeSH Terms: conditions — Obesity | interventions — Blood Specimen Collection; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- assessment of plasmatic lidocaine rate (Experimental): Patients will receive intravenous administration of lidocaine based on a modified body weight ; blood sampling will be performed to assess plasmatic concentration of lidocaine
  Interventions: Biological: Blood sampling; Drug: Lidocaine

INTERVENTIONS:
Biological: Blood sampling
Drug: Lidocaine

SUMMARY:
Intravenous lidocaine is efficient for management of post operative pain in abdominal surgery. As previously published in literature the investigators use it during bariatric surgery.

Nevertheless plasmatic concentration of lidocaine is unknown in this population, despite a widespread use.

Investigators propose in this work to bring an objective proof that administration of lidocaine based on a modified body weight is safe.

Intravenous administration concerned the peri operative period. A total of six samples are taken for each patient.

Investigators get approbation of local ethic committee for this work.

ELIGIBILITY:
Inclusion Criteria:

* Adult who perform a bariatric surgery (sleeve, by-pass, mini by-pass) under laparoscopy
* Body mass index > = 40 kg/m2
* Informed consent signed
* Patient treated with intravenous administration of lidocaine

Exclusion Criteria:

* Contraindication to lidocaine use (allergy, atrioventricular block, seizure, porphyria)
* Concomitant use of beta blocker and others anti arrhythmic drugs
* Cardiac or hepatic insufficiency
* Pregnancy

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Plasmatic concentration of lidocaine | From bolus to day 1 after cessation of administration
  Blood samples will be removed by the peripheral catheter or direct venous puncture with other blood sample usually performed during post-operative period.
  First sample will be taken after initial bolus (ie 10 min after initiation of perfusion), second at 20 min, third at 30 min. The fourth and fifth samples will be taken after change of posology (from 2 to 1 mg/kg/h at the end of surgery) and at the end of administration. The sixth sample will be performed the day after the end of administration.

SECONDARY OUTCOMES:
occurence of adverse events related to lidocaine use | Up to 2 days after surgery
  neurologic (seizure, dysgeusia, dizziness) or cardiologic events (atrio ventricular block, ventricular rhythm disorder) will be assessed after surgery, during hospitalization in post-operative room or intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot - Département d'anesthésie réanimation, Lyon, France

REFERENCES:
- [Result] Carabalona JF, Delwarde B, Duclos A, Le Goff MC, Moulsma M, Citterio-Quentin A, Bouffard Y, Rimmele T. Serum Concentrations of Lidocaine During Bariatric Surgery. Anesth Analg. 2020 Jan;130(1):e5-e8. doi: 10.1213/ANE.0000000000003905. PMID 30399021